CLINICAL TRIAL: NCT01356654
Title: The Use of Transcranial Direct Current Stimulation in the Recovery of Postural Control in Stroke
Brief Title: Transcranial Direct Current Stimulation in Stroke Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Rehabilitation Hospital Hof Ter Schelde (Unknown); Artesis University College, Antwerp (Other)
Responsible Party: Msc Wim Saeys, UZA
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Saeys-1
Record Dates: First submitted 2011-05-10; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Stroke
Keywords: Stroke; TDCS; Gait; Balance; loss of postural balance
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHAM TDCS (Sham Comparator)
  Interventions: Device: Application of Transcranial direct current stimulation (TDCS)
- True TDCS (Active Comparator)
  Interventions: Device: Transcranial Direct current stimulation

INTERVENTIONS:
Device: Application of Transcranial direct current stimulation (TDCS) — Application of TDCS for 20 minutes, 4 times a week for 4 weeks.
  Other Names: tDCS device: CESta, Mind Alive Inc.,Edmonton, Alberta, Canada
  Arms: SHAM TDCS
Device: Transcranial Direct current stimulation — Application of true TDCS for 20min, 4 times a week for 4 weeks.
  Other Names: tDCS device: CESta, Mind Alive Inc., Edmonton, Alberta, Canada
  Arms: True TDCS

SUMMARY:
This study investigates if transcranial Direct Current Stimulation (tDCS) is effective in the recovery of postural control in stroke rehabilitation.

DETAILED DESCRIPTION:
The patients were divided in 2 groups by a randomisation procedure. All patients participated for 2 months in the study. Group 1 received true tDCS in the first month followed by SHAM stimulation in the second month. Group 2 received SHAM in the first month and true stimulation in the following month. Four stimulations of 20minutes were provided during 4 weeks before before changing stimulation intensity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from the consequences of a stroke in the medial cerebral artery, during the sub-acute phase (4-24 weeks after onset)
2. Age between 18-75 years
3. Hospitalised in rehabilitation Hospital Hof Ter Schelde
4. Capable of understanding and giving informed consent

Exclusion Criteria:

1. Cerebellum or brainstem lesions
2. Recently multiple lesions and older lesions which are manifested clinically.
3. History of severe substance abuse (alcohol, drugs, benzodiazepines)
4. Cardiac disease that in the opinion of the clinician precludes participation in the trial (severe dyspnea in rest, severe rhythm disturbances, etc)
5. History of epileptic insults, not caused by the stroke
6. Severe organic co morbidity
7. Psychiatric disorders or history of psychiatric disorders
8. Pace maker / internal defibrillator
9. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale (reporting a change on trunk performance at baseline, after 1 month and after two months) | baseline, after 1 month, After 2 months
  The static sitting balance subscale assesses whether a subject can sit independently and remain seated when the legs are either passively or actively crossed. The dynamic sitting balance subscale evaluates the ability to actively shorten each side of the trunk, first initiated from the shoulder and subsequently initiated from the pelvic girdle. Trunk coordination is evaluated by the possibility to independently rotate the upper and lower part of the trunk. The scoring range for the static and dynamic sitting balance and coordination subscales are 7, 10 and 6 points respectively.
Rivermead Motor Assessment Battery (RMAB) (reporting a change on motricity of gross function, arm, leg and trunk at baseline, after 1 month and after two months) | baseline, after 1 month, After 2 months
  The RMAB assesses the motor performance of patients with stroke.32 It consists of test items clustered in three sections that are ordered hierarchically. The gross function subscale (13 items), the Leg and Trunk subscale (10 items) and the arm subscale (15 items)
Tinetti Test (reporting a change on balance and gait tasks at baseline, after 1 month and after two months) | baseline, after 1 month, After 2 months
  The Tinetti Test is an easily performed test that measures a patients' gait and balance. The individual scores are combined to form three measures; a gait score, a standing balance score and a total score.
  The maximum score for the gait component and the balance component are 12 and 16 points respectively, resulting in a maximum of 28 points for the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital Hof Ter Schelde, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411